CLINICAL TRIAL: NCT02193451
Title: Urodynamics for Prostate Surgery Trial; Randomised Evaluation of Assessment Methods (UPSTREAM) for Diagnosis and Management of Bladder Outlet Obstruction in Men
Brief Title: Urodynamics for Prostate Surgery Trial; Randomised Evaluation of Assessment Methods
Acronym: UPSTREAM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: North Bristol NHS Trust (Other)
Collaborators: University of Bristol (Other); University of Aberdeen (Other); Newcastle University (Other); Royal Devon and Exeter NHS Foundation Trust (Other); University of Sheffield (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: UPSTREAM 3250; 12/140/01 (Other Grant/Funding Number: NIHR HTA)
Record Dates: First submitted 2014-07-16; First posted 2014-07-17 (Estimated); Last update posted 2020-01-10 (Actual); Status verified 2019-12

CONDITIONS: Lower Urinary Tract Symptoms; Voiding Dysfunction; Benign Prostate Obstruction; Detrusor Underactivity
Keywords: Lower urinary tract symptoms; Male LUTS; Voiding dysfunction; Benign prostate obstruction; Detrusor underactivity
MeSH Terms: conditions — Lower Urinary Tract Symptoms; Urinary Bladder, Underactive | interventions — Urodynamics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Urodynamics (Experimental): Invasive urodynamic cystometry including pressure flow studies, along with usual diagnostics in male LUTS
  Interventions: Procedure: Urodynamics; Procedure: Usual care
- Usual care (Active Comparator): Usual diagnostics in male LUTS; flow rate test, symptom score and bladder diary
  Interventions: Procedure: Usual care

INTERVENTIONS:
Procedure: Urodynamics — Diagnostic test for urinary storage and voiding function
  Other Names: Cystometry; Pressure flow study
  Arms: Urodynamics
Procedure: Usual care
  Other Names: Flow rate; Symptom scores; Bladder diary

SUMMARY:
Background and study aims: The prostate gland sits around the exit of the bladder in men. As men get older, the prostate grows, and this can narrow the exit from the bladder, so that there is restriction of flow. As a result, some men develop difficulty passing urine (voiding) as they age. For these men, prostate surgery can be helpful by removing the part of the prostate causing the narrowing, so that flow improves. However, for some men, almost identical symptoms of difficulty passing urine are due to underactive bladder. In other words, the bladder contraction is too weak, and is not effective at expelling the urine. This is a smaller group, but important, as these men may have no improvement after prostate surgery, while being exposed to risk of complications of surgery. Medical assessment of men with voiding problems typically involves discussing the symptoms, doing a physical examination of the prostate and measuring the urine flow rate. In many NHS hospitals, these are the only tests done before deciding whether to proceed to prostate surgery. In effect, voiding symptoms are presumed to be a result of prostate enlargement for these men, since it is the more common problem compared with bladder underactivity. However, this approach cannot identify which men actually have bladder underactivity as the cause of their voiding symptoms. So, in some hospitals an extra test is used, called urodynamics. Urodynamics is done to measure how much pressure the bladder generates when passing urine, because a high pressure shows the problem is obstruction, and a low pressure shows it is bladder weakness. Urodynamics involves gently putting a small tube into the bladder via the penis to measure the bladder pressure, and to fill the bladder with a sterile fluid (saline). Another small tube is gently placed into the rectum, via the anus, to measure abdominal pressures. Measuring abdominal pressure is necessary because any change in abdominal pressure can affect bladder pressure, and if the test did not allow for this it could give a misleading result. Urodynamics is safe, but some men find it uncomfortable or undignified, and a few develop urine infection afterwards. No studies have been conducted so far to tell us which of these two approaches to assessing men with voiding urinary problems is better overall.

UPSTREAM consists of two phases: "UPSTREAM - Phase I" was a pragmatic, two-arm, multicentre, randomised controlled trial (RCT) to determine the clinical and cost-effectiveness of invasive urodynamics (UDS) for the diagnosis and management of bladder outlet obstruction in men. Men from 26 urology departments of NHS Hospitals in England who had bothersome lower urinary tract symptoms (LUTS) and were seeking further treatment, which may have included surgery, were randomised to one of two study arms; 'Routine Care' (as per the NICE diagnostic pathway), or routine care plus UDS ('Urodynamics'), which is currently optional. The design was utilised to establish noninferiority in symptom severity (International Prostate Symptom Score [IPSS]) 18-months post-randomisation. The primary outcome was IPSS at 18-months post-randomisation, and a key secondary outcome was the influence of UDS on rates of bladder outlet surgery. The RCT started 01 April 2014 and ended 30 September 2018.

In 2018, we were awarded an extension to conduct a further (long term) follow up of UPSTREAM participants, five years post-randomisation; "UPSTREAM - Phase II". We aim to identify: the symptom outcomes of treatment; definitive surgery rates in the two study arms; and the long-term impact of LUTS and its therapy. The focus will continue to be on effectiveness and patient outcomes as per the original commissioning brief. "UPSTREAM - Phase II" started 01 July 2019 and has a planned end date of 30 June 2022.

DETAILED DESCRIPTION:
The aim of the UPSTREAM trial ("UPSTREAM - Phase I") was to determine whether a care pathway including invasive urodynamics is no worse for men in terms of symptom outcome than one in which it is not included, at 18 months after randomisation. We also aimed to establish whether inclusion of invasive urodynamics reduces rates of bladder outlet surgery as a main secondary outcome.

The following men were invited to participate (inclusion criterion); • Men seeking further treatment for their bothersome lower urinary tract symptoms (LUTS) which may include surgery

Men were not invited to participate (exclusion criteria) if they:

* were unable to pass urine without a catheter (urinary retention)
* had a relevant neurological disease, such as a stroke
* were undergoing treatment for prostate or bladder cancer
* had previously had prostate surgery
* were not medically fit for surgery, or were unable to complete outcome assessments
* did not consent to be assigned at random to one of the pathways

We compared the two methods of investigation by finding out whether the men had similar relief of their symptoms, by measuring the change in the prostate symptom score (IPSS) in the two groups at 18 months after randomisation (primary outcome).

We also looked at the following secondary outcomes:

* Whether the invasive tests changed the decision for surgery in some of the men (how many men had surgery in each of the two groups?)
* The cost-effectiveness of the two management pathways
* Adverse effects of (a) the tests and (b) the treatments (e.g. urinary infection, urinary retention)
* Urinary symptoms at 6, 12 & 18 months, using the International Consultation on Incontinence Questionnaires (ICIQ) and the Male Lower Urinary Tract Symptoms questionnaire (ICIQ-MLUTS)
* Quality of life, using the IPSS-QoL question
* Sexual function, using the ICIQ-MLUTS sex questionnaire
* Satisfaction with urodynamic testing, using the ICIQ-UDS-S questionnaire
* The maximum urinary flow rate (Qmax) at 18 months
* Health outcomes, using the EQ-5D-5L questionnaire

For "UPSTREAM - Phase II". In this further follow up study ("UPSTREAM - Phase II"), we want to find out the longer term (5-year) results of treatment for the men's LUTS, and see how many men went on to receive surgery after the initial 18-months (i.e. after the original study, "UPSTREAM - Phase I").

We will approach existing participants of the UPSTREAM trial ("UPSTREAM - Phase I"). In taking part in "UPSTREAM - Phase II", men do not need to return to hospital for any clinical assessments. Instead we will ask them to complete one questionnaire booklet about their urinary symptoms, the effect on their everyday life, and their general state of health. We will also securely collect information relevant to this study from central NHS records (such as information about relevant inpatient stays and outpatient attendances).

Outcome measures will include:

LUTS will be measured with the widely-used patient reported outcome, the International Prostate Symptom Score (IPSS), at five years post-randomisation.

• Measures from the International Consultation on Incontinence Questionnaires (ICIQ) will also be used, giving sensitive and comprehensive assessment of LUTS severity/ bother, sexual function and quality of life (QoL), i.e.: O IPSS QoL O ICIQ Male LUTS (ICIQ-MLUTS) O ICIQ sexual function in Male LUTS (ICIQ-MLUTS-sex)

* The EQ-5D-5L will be used to provide the QoL weights used to calculate Quality Adjusted Life Years (QALYs).
* Data for: Surgery rates (the relative proportion of men in each group having surgery up to five years post-randomisation); diagnostic testing after the main trial (where possible); and resource use will be obtained via a one-off bespoke data extraction of Health Episode Statistics (HES) and HES-Office of National Statistics (ONS) linked data, via NHS Digital. This will include individual level data about participants' relevant: inpatient stays; outpatient attendances: including procedures; radiology and accident and emergency (A&E) episodes; and cause of death (where applicable).

ELIGIBILITY:
"UPSTREAM - Phase I":

Inclusion Criteria:

* Men seeking further treatment for their bothersome lower urinary tract symptoms (LUTS) which may include surgery

Exclusion Criteria:

* unable to pass urine without a catheter (urinary retention)
* relevant neurological disease, such as a stroke
* undergoing treatment for prostate or bladder cancer
* previously had prostate surgery
* not medically fit for surgery, or are unable to complete outcome assessments
* do not consent to be assigned at random to one of the pathways

"UPSTREAM - Phase II":

Inclusion criteria:

PROMS (questionnaire) study component:

Men randomised (enrolled) to the UPSTREAM trial (Phase I) who were willing to be contacted for long term follow up, as indicated on their original (Phase I) consent form.

NHS Digital data extraction study component:

Men randomised (enrolled) to the UPSTREAM trial (Phase I).

Exclusion criteria:

PROMS (questionnaire) study component:

1. Patients who are not already randomised (enrolled) to the UPSTREAM trial (Phase I)
2. UPSTREAM (Phase I) participants who:

2.1. are not willing to be contacted about long term follow up 2.2. have withdrawn trial participation, or at least withdrawn permission to be contacted in the future for long term follow up, at the time of their 18-month timepoint 2.3. do not consent and/or are not willing or able to comply with essential study procedures of this further follow up (UPSTREAM - Phase II)

NHS Digital data extraction study component:

1. Patients who are not already randomised (enrolled) to the UPSTREAM trial (Phase I)
2. UPSTREAM (Phase I) participants who have withdrawn permission for the study to continue to access sections of their medical notes and NHS records, ONS and NHS Central registers information, at the time of their 18-month timepoint

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 820 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
International Prostate Symptom Score | 18 months
  Primary clinical outcome: difference in lower urinary tract symptom (LUTS) between the two arms at 18 months, measured with the International Prostate Symptom Score (IPSS)

SECONDARY OUTCOMES:
Surgery rate | 18 months
  The relative proportion of men in each group having surgery up to 18 months after randomisation
Cost-effectiveness analyses | 18 months
  Cost effectiveness from the perspectives of the Health Service, Personal Social Services and patients
Adverse events | 18 months
  Adverse events of testing and treatment (e.g. infection, urinary retention).
International Consultation on Incontinence Questionnaires | 18 months
  Measures from the International Consultation on Incontinence Questionnaires (ICIQ) regarding LUTS severity/ bother, sexual function, quality of life and satisfaction with urodynamic testing. The following will be measured at 6, 12 and 18 months; IPSS (including quality of life) ICIQ Male LUTS (ICIQ-MLUTS) ICIQ sexual function in Male LUTS (ICIQ-MLUTS-sex)
Maximum urinary flow rate | 18 months
  Maximum urinary flow rate (Qmax) at 18 months. In men undergoing surgery in both arms, an additional Qmax measure at 4 months after operation will be used as a quality measure for surgery.
EQ-5D-5L | 18 months
  EQ-5D-5L consists of the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). In the descriptive system, respondents rate their health 'TODAY' according to 5 dimensions (Mobility; Self-Care; Usual Activities; Pain/Discomfort; and Anxiety/Depression), with 5 levels of severity (No Problems; Slight; Moderate; Severe; and Extreme Problems). This results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions are combined into a 5-digit number that describes the patient's health state. The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' (100) and 'The worst health you can imagine' (0). The VAS can be used as a quantitative measure of health outcome reflecting the patient's own judgement. Full details of the scoring system can be found via the EQ-5D website/user guide.
International Prostate Symptom Score (IPSS) | 5 years post randomisation ("UPSTREAM - Phase II")
  "UPSTREAM - Phase II": difference in lower urinary tract symptom (LUTS)
Surgery rate | 5 years post randomisation ("UPSTREAM - Phase II")
  "UPSTREAM - Phase II": The relative proportion of men in each group having surgery up to 5 years after randomisation
Measures from the International Consultation on Incontinence Questionnaires (ICIQ) regarding male lower urinary tract symptoms (LUTS) severity/ bother | 5 years post randomisation ("UPSTREAM - Phase II")
  "UPSTREAM - Phase II": ICIQ Male LUTS (ICIQ-MLUTS); questionnaire evaluating MLUTS and impact on quality of life. 13 items, Scoring: 0-20 voiding symptoms subscale 0-24 incontinence symptoms subscale. Bother scales are not incorporated in the overall score but indicate impact of individual symptoms for the patient. See https://iciq.net for further information.
Measures from the International Consultation on Incontinence Questionnaires Measures from the International Consultation on Incontinence Questionnaires (ICIQ) regarding regarding sexual function | 5 years post randomisation ("UPSTREAM - Phase II")
  "UPSTREAM - Phase II":ICIQ sexual function in Male LUTS (ICIQ-MLUTS-sex). Patient-complete questionnaire for evaluation of male sexual function associated with their MLUTS and impact of quality of life. 4 items, scoring: 0-12 overall score with greater values indicating increasing problems with sexual matters. Bother scales are not incorporated in the overall score but indicate impact of individual symptoms for the patient. See https://iciq.net for further information.
Quality of Life (QoL) | 5 years post randomisation ("UPSTREAM - Phase II")
  "UPSTREAM - Phase II": International Prostate Symptom Score (IPSS) including QoL question. The IPSS is based on the answers to seven questions concerning urinary symptoms and one question concerning quality of life. Each question concerning urinary symptoms allows the patient to choose one out of six answers indicating increasing severity of the particular symptom. The answers are assigned points from 0 to 5. The total score can therefore range from 0 to 35 (asymptomatic to very symptomatic).
EQ-5D-5L | 5 years post randomisation ("UPSTREAM - Phase II")
  "UPSTREAM - Phase II": EQ-5D-5L consists of the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). In the descriptive system, respondents rate their health 'TODAY' according to 5 dimensions (Mobility; Self-Care; Usual Activities; Pain/Discomfort; and Anxiety/Depression), with 5 levels of severity (No Problems; Slight; Moderate; Severe; and Extreme Problems). This results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions are combined into a 5-digit number that describes the patient's health state. The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' (100) and 'The worst health you can imagine' (0). The VAS can be used as a quantitative measure of health outcome reflecting the patient's own judgement. Full details of the scoring system can be found via the EQ-5D website/user guide.

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Drake, DM, MA, FRCS(Urol), Principal Investigator — University of Bristol; Athene Lane, PhD, Study Director — University of Bristol
Locations (1):
- North Bristol NHS Trust, Bristol, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Young GJ, Lewis AL, Lane JA, Winton HL, Drake MJ, Blair PS. Statistical analysis plan for the Urodynamics for Prostate Surgery Trial; Randomised Evaluation of Assessment Methods (UPSTREAM). Trials. 2017 Oct 3;18(1):455. doi: 10.1186/s13063-017-2206-y. PMID 28974250
- [Background] Bailey K, Abrams P, Blair PS, Chapple C, Glazener C, Horwood J, Lane JA, McGrath J, Noble S, Pickard R, Taylor G, Young GJ, Drake MJ, Lewis AL. Urodynamics for Prostate Surgery Trial; Randomised Evaluation of Assessment Methods (UPSTREAM) for diagnosis and management of bladder outlet obstruction in men: study protocol for a randomised controlled trial. Trials. 2015 Dec 10;16:567. doi: 10.1186/s13063-015-1087-1. PMID 26651344
- [Background] Drake MJ, Lewis AL, Lane JA. Urodynamic Testing for Men with Voiding Symptoms Considering Interventional Therapy: The Merits of a Properly Constructed Randomised Trial. Eur Urol. 2016 May;69(5):759-60. doi: 10.1016/j.eururo.2016.01.035. Epub 2016 Feb 1. PMID 26847139
- [Result] Selman LE, Ochieng CA, Lewis AL, Drake MJ, Horwood J. Recommendations for conducting invasive urodynamics for men with lower urinary tract symptoms: Qualitative interview findings from a large randomized controlled trial (UPSTREAM). Neurourol Urodyn. 2019 Jan;38(1):320-329. doi: 10.1002/nau.23855. Epub 2018 Oct 12. PMID 30311686
- [Result] Lewis AL, Young GJ, Abrams P, Blair PS, Chapple C, Glazener CMA, Horwood J, McGrath JS, Noble S, Taylor GT, Ito H, Belal M, Davies MC, Dickinson AJ, Foley CL, Foley S, Fulford S, Gammal MM, Garthwaite M, Harris MRE, Ilie PC, Jones R, Sabbagh S, Mason RG, McLarty E, Mishra V, Mom J, Morley R, Natale S, Nitkunan T, Page T, Payne D, Rashid TG, Saeb-Parsy K, Sandhu SS, Simoes A, Singh G, Sullivan M, Tempest HV, Viswanath S, Walker RMH, Lane JA, Drake MJ. Clinical and Patient-reported Outcome Measures in Men Referred for Consideration of Surgery to Treat Lower Urinary Tract Symptoms: Baseline Results and Diagnostic Findings of the Urodynamics for Prostate Surgery Trial; Randomised Evaluation of Assessment Methods (UPSTREAM). Eur Urol Focus. 2019 May;5(3):340-350. doi: 10.1016/j.euf.2019.04.006. Epub 2019 Apr 30. PMID 31047905
- [Derived] Wei DY, Drake MJ. Undiagnosed neurological disease as a potential cause of male lower urinary tract symptoms. Curr Opin Urol. 2016 Jan;26(1):11-6. doi: 10.1097/MOU.0000000000000243. PMID 26555692